CLINICAL TRIAL: NCT04337333
Title: Feasibility and Safety of a Newly Developed Two-in-one Covered and Uncovered Metal Stent for Inoperable Malignant Distal Biliary Obstruction
Brief Title: Two-in-one Covered and Uncovered Metal Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jin Hong Kim, Professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-DEV-INT-20-035
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Extrahepatic Bile Duct Cancer; Pancreatic Cancer; Lymph Node Metastases; Gallbladder Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Pancreatic Neoplasms; Lymphatic Metastasis; Gallbladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two-in-one stent (Other): Endoscopic placement of a Two-in-one stent into the extrahepatic bile duct, considering the longitudinal location of the stricture segment and predicted safety margin
  Interventions: Device: Two-in-one stent

INTERVENTIONS:
Device: Two-in-one stent — Endoscopic placement of a Two-in-one metal stent into extrahepatic bile duct

SUMMARY:
Endoscopic placement of a self-expandable metal stent (SEMS) is the principle method for palliation of inoperable malignant distal biliary obstruction. However, none of bare, covered, and anti-reflux metal stent alone constantly demonstrated superiority over the others in the stent patency. To compensate for the limitations of each stent, a double stent system in which both covered and bare SEMSs are integrated into one stent system was introduced. In the current study, the investigators aimed to evaluate the efficacy and safety of this stent in patients with inoperable malignant distal biliary obstruction.

DETAILED DESCRIPTION:
Endoscopic placement of a self-expandable metal stent (SEMS) is the principle method for palliation of inoperable malignant distal biliary obstruction. As the survival time for those patients has improved due mainly in part to development of chemotherapeutic intervention, it is becoming important to prevent recurrent cholangitis and liver failure by prolonging the SEMS patency, leading to continuation of chemotherapy and better prognosis. Therefore, one-time stent insertion before disease-progression-related death is an ultimate goal of developing an ideal biliary stent.

SEMSs have been found to be superior to plastic stents in terms of the stent patency, because it prevent accumulation of biliary sludge owing to larger diameter. The ideal designs of biliary SEMSs for prolongation of the stent patency include 1) bare metal mesh for tissue embedding to prevent stent migration, 2) covering material to counteract neoplastic tumor ingrowth, and 3) anti-reflux structure to reduce enteric biliary reflux. However, none of bare, covered, and anti-reflux metal stent alone constantly demonstrated superiority over the others in the stent patency.

To compensate for the limitations of each stent, a double stent system in which both covered and bare SEMSs are integrated into one stent system was introduced in the field of the interventional radiology, but further data accumulation is needed to assess the comparability with various conventional SEMS types in terms of stent patency, reintervention efficacy, and clinical outcomes following reintervention, because in this system two metal stents are implanted at once exclusively via percutaneous route and clogged inner covered stent cannot be removed at the time of the reintervention. Recently a new covered and uncovered SEMS in which the clogged inner stent can be endoscopically removed leaving the outer stent in place, was introduced. In the current study, we aimed to evaluate the efficacy and safety of this stent in patients with inoperable malignant distal biliary obstruction.

ELIGIBILITY:
Inclusion Criteria:

ㆍMalignant biliary obstruction, 2 cm distal to the hilum ㆍNot eligible for curative surgical resection owing to metastasis, locally advanced stage, or high operation risk ㆍEastern Cooperative Oncology Group Performance status 0-3

Exclusion Criteria:

ㆍBeing evaluated for potential benign biliary stricture or possible operation ㆍHistory of biliary surgery except cholecystectomy ㆍCoagulopathy (International normalized ratio >1.5, platelet count <50,000) ㆍCoexist other organ dysfunction (American Society of Anesthesiologist physical status grade III or IV) ㆍInability to obtain informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative patency of inner covered stent and Two-in-one stent | From the date of stent insertion until the date of first documented stent dysfunction, assessed upto 12 months

SECONDARY OUTCOMES:
Overall patient survival | From the date of stent insertion until the date of death from any cause, assessed upto 12 months
Stent dysfunction-free patient survival | From the date of stent insertion until the date of first documented stent dysfunction or the date of death from any cause, whichever came first, assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hong Kim, MD, PhD, Study Director — Ajou University School of Medicine
Locations (2):
- South Korea (2):
  - Ajou University Hospital, Suwon, Gyeong Gi Do
  - Ajou University Hospital, Suwon, Gyeonggido

IPD SHARING:
Plan to Share IPD: No